CLINICAL TRIAL: NCT05967715
Title: Exercise Training Influences Gut Microbiota and Cardiovascular Health Through Inflammation Control in Adult Hypertensive Population: the MicroFit Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Collaborators: Actial Farmaceutica S.r.l. (Industry)
Responsible Party: Principal Investigator, Davide Agnoletti, Assistant Professor, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MicroFit
Record Dates: First submitted 2023-06-16; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Hypertension; Microbiota
Keywords: hypertension; gut microbiota; exercise training; physical activity; central hemodynamics; arterial stiffness; pulse wave velocity
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Exercise; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only for the "probiotics" and "placebo" arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise training (Experimental): high intensity interval training: thrice a week
  Interventions: Behavioral: exercise training
- Probiotics (Active Comparator): VSL#3# probiotic: twice daily
  Interventions: Other: Probiotics
- Placebo (Placebo Comparator): Comparator of the Probiotics arm
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: exercise training — high intensity interval training
  Arms: Exercise training
Other: Probiotics — VSL#3# Probiotic
  Arms: Probiotics
Other: Placebo — Probiotic Placebo
  Arms: Placebo

SUMMARY:
Cardiovascular diseases are the number 1 cause of death globally, taking an estimated 17.9 million lives each year (31% of deaths worldwide). Hypertension, with 1.13 billion people affected worldwide, is the leading risk factor for global mortality. Physical inactivity is among the modifiable cardiovascular risk factors. While the beneficial effects of physical activity on cardiovascular system are widely known, the mechanisms involved are not completely understood. Both exercise training and hypertension are linked to inflammation. Furthermore, there is evidence that gut microbiota regulates inflammatory patterns. Recent investigations showed a relationship between exercise training and the composition/functionality of the gut microbiota. Anyway, the modification of the composition and functionality of the gut microbiota in hypertension due to the exercise training and the relative involvement of oxidative stress and inflammation are not completely understood.

In literature an association between gut microbiota composition and arterial stiffness is described, in particular, the investigators observed both a direct correlation between arterial stiffness and abundances of bacteria associated with altered gut permeability and inflammation; and an inverse relationship between arterial stiffness, microbiota diversity, and abundances of bacteria associated with most fit microbiota composition. Anyway, while these association were stable in animal studies, in human studies none of the identified interventional trials was able to demonstrate this relationship. Of note, only half of human studies measured BP, and very few adjusted the vascular analyses for BP variation, which is a major determinant of arterial stiffness.

This is a non-profit, monocentric, non-pharmacological interventional study, a randomized controlled trial with three intervention arms, partial double-blind, aiming to verify the hypothesis that, in hypertensive patients in primary prevention with cardiovascular risk factors, physical exercise favorably modifies the intestinal bacterial flora compared to the probiotic, with a positive impact on cardiovascular health, and to demonstrate that this involves inflammation modulation. There will be 3 intervention arms, with 1:1:1 stratified randomization by gender: 1. Administration of controlled physical activity training; 2. Administration of probiotic; 3. Administration of placebo. Arms 2 and 3 will be double-blind. The intervention will last for three months, followed by a 6-month follow-up period. Afterwards, the medical team may be contacted for further tests/assessments or simply for information about the participant's health status, for a total duration of 24 months.

The investigators hypothesize that hypertensive patients in cardiovascular primary prevention have a dysbiotic gut microbial signatures, that could be a new marker of early vascular aging. Secondly, the investigators anticipate that exercise training will modify both gut microbiota and hemodynamic profile, and that a relationship exists between gut microbiota and hemodynamic modifications. Thirdly, the investigators expect that the beneficial effects of exercise training are driven by positive changes in the inflammatory modulators.

ELIGIBILITY:
Inclusion Criteria:

* Arterial hypertension*;
* Stable antihypertensive therapy in the last 2 months, with controlled blood pressure values;
* Age 40-65 years;
* Willing to sign the written informed consent;
* Written and spoken Italian language comprehension.

Exclusion Criteria:

* Atrial fibrillation;
* Diabetes mellitus either type I or II;
* Active cancer;
* Inflammatory bowel disease;
* Heart failure NYHA class III to IV;
* Recent antibiotic or probiotic treatment in the previous month for any reason;
* Recent myocardial infarction or hospital admission for any other reason in the previous 6 months;
* Any other condition that the medical doctor (MD) considers to contraindicate the participation in an exercise program of High intensity;
* Pulmonary disease requiring oxygen therapy;
* Relevant neurological condition impairing motor or cognitive function;
* Severe depressive disorder;
* Pregnancy.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-04-02 (Estimated); Study Completion 2026-04-02 (Estimated)

PRIMARY OUTCOMES:
To describe the modification of the gut microbiota composition and function after the exercise training compared to probiotic supplements and to placebo. | time 0 and 3 months
  Changes in measures of gut microbiota composition and function from time 0 to 3 months (alpha diversity, beta diversity, taxonomy, relative abundance of microbial genes and pathways)

SECONDARY OUTCOMES:
To describe the association between gut microbiota patterns with impaired central hemodynamics | time 0 and 3 months
  To measure the association of gut microbiota diversity indexes, taxonomy, relative abundance of microbial genes and pathways, with central hemodynamics parameters (central blood pressure, aortic stiffness, pulse pressure amplification, augmentation index).
To test the association of the systemic inflammation with the modification of gut microbiota composition/functionality. | time 0 and 3 months
  To test the association between inflammatory markers (alpha-1-acid glycoprotein, high-sensitive c-reactive protein) and gut microbiota diversity indexes, taxonomy, relative abundance of microbial genes and pathways.
To test the modification of endothelial function after the exercise training in comparison to probiotic supplements and placebo. | time 0, and 3 months
  To measure variation in endothelial glycocalyx thickness before and after 3-mo intervention
To identify the variation of the gut microbiota composition and function in the long term follow up after the intervention | from 3 to 9 months.
  Measures of gut microbiota diversity indexes, taxonomy, relative abundance of microbial genes and pathways at the end of the intervention (3 months) and after the 9-mo follow up.
To describe the association between gut microbiota patterns with impaired central hemodynamics in the long term follow up 6 months after the intervention | at 9-mo follow up
  To measure the association of gut microbiota diversity indexes, taxonomy, relative abundance of microbial genes and pathways, with central hemodynamics parameters (central blood pressure, aortic stiffness, pulse pressure amplification, augmentation index)
To test the association of the systemic inflammation with the modification of gut microbiota composition/functionality, after the long term follow up 6 months after the intervention. | at 9-mo follow up
  To test the association between inflammatory markers (alpha-1-acid glycoprotein, high-sensitive c-reactive protein) and gut microbiota diversity indexes, taxonomy, relative abundance of microbial genes and pathways, at 9-mo follow up.
To test the modification of endothelial function after the exercise training in comparison to probiotic supplements and placebo, after the long term follow up 6 months after the intervention | at 9-mo follow up
  To measure variation in endothelial glycocalyx thickness at 9-mo follow up

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No